CLINICAL TRIAL: NCT00331864
Title: A Phase IIIb, Open-label, Multi-center 12 Month Study to Evaluate the Safety, Tolerability and Efficacy of Ranibizumab (0.3 mg and/or 0.5 mg) in Patients With Subfoveal Choroidal Neovasculariza-tion Secondary to Age-related Macular Degeneration
Brief Title: SUSTAIN - Study of Ranibizumab in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-Related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002A2303
Record Dates: First submitted 2006-04-11; First posted 2006-05-31 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization
Keywords: AMD, ranibizumab
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

ARMS (1):
- Ranibizumab (Experimental): Ranibizumab-naïve (Non-ANCHOR) patients received up to 12 intravitreal injections (Month 0 through Month 11). The dose of 0.3 mg ranibizumab was administered monthly for three consecutive months. From Month 3 through Month 11, either 0.3 mg ranibizumab or, after implementation of an amendment to the protocol, 0.5 mg ranibizumab were injected as individually needed based on re-treatment criteria described in the protocol. For patients who had participated in the ANCHOR study, either 0.3 mg ranibizumab or, after implementation of an amendment to the protocol, 0.5 mg ranibizumab was injected if the patient met re-treatment criteria described in the protocol. Ranibizumab was administered no sooner than 14 days after the previous treatment.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab
  Other Names: rhuFab V2

SUMMARY:
Ranibizumab is a humanised recombinant monoclonal antibody fragment targeted against human vascular endothelial growth factor A. This study will assess the safety and efficacy of ranibizumab administered on an as-needed dosing regimen in patients with subfoveal choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Patients who participated in this study included those who had completed participation in the study CRFB002A2301 (ANCHOR; NCT00061594), newly diagnosed patients, as well as previously diagnosed patients who had had recent disease progression.

Inclusion Criteria:

* Male or female patients > 50 years of age
* Diagnosis of active primary or recurrent CNV secondary to AMD, including those with predominantly classic, minimally classic or occult lesions with no classic component
* The total area of CNV (including both classic and occult components) encompassed within the lesion must be >= 50% of the total lesion area
* The total lesion area must be <= 12 disc areas
* Patients who have a BCVA (best corrected visual acuity) score between 73 and 24 letters, inclusive, in the study eye using ETDRS-like (Early Treatment of Diabetic Retinopathy Study) grading charts (approximately 20/40 to 20/320)

Exclusion Criteria:

* Patients who have a BCVA of < 34 letters in both eyes (legally blind is defined as bilateral vision below 20/200 or less than 34 letters)
* Laser photocoagulation, treatment with intravitreal steroids, verteporfin photo dynamic therapy or pegaptanib sodium in the study eye within 30 days preceding Day 1
* Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, protein kinase C inhibitors, etc.)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Customer Information, Study Chair — Novartis - Including Sites in Germany
Locations (1):
- Novartis - 64 sites in 11 countries, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of two groups, one group being naïve to ranibizumab ("Non-ANCHOR" patients) and the other group were those patients who previously were treated with ranibizumab in the ANCHOR study (NCT00061594; "ANCHOR" patients).
Groups:
- Ranibizumab Non-ANCHOR: Patients received up to 12 intravitreal injections (Month 0 through Month 11). The dose of 0.3 mg ranibizumab was administered monthly for three consecutive months. From Month 3 through Month 11, either 0.3 mg ranibizumab or, after implementation of an amendment to the protocol, 0.5 mg ranibizumab were injected as individually needed based on retreatment criteria described in the protocol. Ranibizumab was administered no sooner than 14 days after the previous treatment.
- Ranibizumab ANCHOR: Patients received up to 12 intravitreal injections (Month 0 through Month 11). From Month 0 through Month 11, either 0.3 mg ranibizumab or, after implementation of an amendment to the protocol, 0.5 mg ranibizumab was injected if the patient met retreatment criteria described in the protocol. Ranibizumab was administered no sooner than 14 days after the previous treatment.
Period: Overall Study
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Started | 513 | 18
Completed | 455 | 14
Not Completed | 58 | 4
Not completed — Adverse Event | 30 | 1
Not completed — Lack of Efficacy | 4 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 10 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Administrative Problems | 1 | 0
Not completed — Death | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR | Total
Number analyzed (Participants) | 513 | 18 | 531
Age, Customized [Number; unit: participants]
  < 50 years | 1 | 0 | 1
  50 to < 65 years | 49 | 0 | 49
  65 to < 75 years | 173 | 5 | 178
  75 to < 85 years | 230 | 12 | 242
  ≥ 85 years | 60 | 1 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 9 | 303
  Male | 219 | 9 | 228

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Ocular Adverse Events (AEs) in the Study Eye
Description: Percentage of patients with ocular adverse events in the study eye over the one year (12 month) treatment period.
Time Frame: Baseline through end of study (12 month treatment period)
Population: For Non-ANCHOR treatment group, the analysis population was the Safety population: All patients who had received at least one application of study drug and had at least one post-baseline safety assessment. For the ANCHOR treatment group, the analysis population was all enrolled patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 513 | 18
Percentage of Participants | 48.5 | 38.9

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) of the Study Eye From Baseline to Month 3
Description: BCVA was assessed using best correction determined from protocol refraction. BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts at an initial testing distance of 4 meters.
  BCVA is measured by the number of letters a patient could correctly read on an eye chart; hence an increased score indicates improvement in acuity.
Time Frame: Baseline and Month 3
Population: Non-ANCHOR patients: Analysis of Intent-to-Treat (ITT) population (all patients who received study drug at least once and had at least one post-baseline efficacy assessment) using last observation carried forward (LOCF). ANCHOR patients: Analysis of All Enrolled population (all enrolled patients) using LOCF.
Measure: Mean (Standard Deviation); unit: Letters on the ETDRS-like testing charts
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 509 | 15
Letters on the ETDRS-like testing charts
  Baseline | 56.2 (12.11) | 47.2 (22.10)
  Change to Month 3 | 5.8 (11.12) | 1.9 (9.26)

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) of the Study Eye From Baseline to Month 12
Description: as for outcome 2
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Letters on the ETDRS-like testing charts
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 509 | 17
Letters on the ETDRS-like testing charts
  Baseline | 56.2 (12.11) | 47.2 (22.10)
  Change to Month 12 | 3.6 (13.89) | 1.6 (8.66)

4. Secondary Outcome: Mean Change in Central Retinal Thickness of the Study Eye From Baseline to Month 3
Description: Central retinal thickness was assessed using optical coherence tomography (OCT). OCT imaging was performed by trained personnel at each site using the Zeiss Stratus OCT™ 3 with version A6.1 (or more recent) software. Analysis of the OCT images was performed by the investigator. A negative number indicates improvement (reduced thickness).
Time Frame: Baseline and Month 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrometers
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 507 | 15
Micrometers
  Baseline | 339.6 (109.38) | 214.1 (64.92)
  Change to Month 3 | -101.1 (115.69) | 36.3 (72.96)

5. Secondary Outcome: Mean Change in Central Retinal Thickness of the Study Eye From Baseline to Month 12
Description: as for outcome 4
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrometers
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 507 | 17
Micrometers
  Baseline | 339.6 (109.38) | 214.1 (64.92)
  Change to Month 12 | -91.5 (115.47) | 39.3 (84.61)

6. Secondary Outcome: Time to the First Retreatment After Month 2
Description: Time to first re-treatment is calculated as time difference in months starting from Month 2 until the month of first re-treatment.
  Criteria for re-treatment:
  * a >5 letter decrease in BCVA (determined using EDRS charts) based upon the highest visual acuity score from any prior scheduled study visit (Months 0, 1, 2 or 3)
  * a >100 µm increase in central retinal thickness (determined using OCT) from the thinnest measurement from any prior scheduled study visit (Months 0, 1, 2 or 3)
Time Frame: Month 2 to Month 11
Population: Intent-to-Treat (ITT) population patients: All patients who received study drug at least once and had at least one post-baseline efficacy assessment. The ANCHOR patients were not included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Ranibizumab Non-ANCHOR
Number analyzed (Participants) | 500
Months | 2 [1 to 6]

7. Secondary Outcome: Total Number of Treatments
Description: Total number of treatments administered during the entire treatment period (Month 0 to 11).
Time Frame: Baseline (Month 0) to Month 11
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Treatments
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 513 | 18
Treatments | 5.6 (2.37) | 1.1 (2.29)

8. Primary Outcome: Percentage of Patients With Targeted Grade 3 Adverse Events (AEs) in the Study Eye
Description: Grade 3 targeted AEs included:
  * 4+ ocular inflammation or 2-3+ ocular inflammation failing to decrease to ≤ 1+ within 30 days
  * ≥ 30 letter decrease in BCVA that developed within 14 days of ranibizumab injection
  * sustained (>15 minutes) loss of light perception due to elevated intraocular pressure (IOP) or a >20 mm Hg change in IOP persisting longer than 14 days
  * new retinal tear or detachment involving the macula
  * new vitreous hemorrhage >2+ severity not resolving within 14 days
  * new or increase of previous retinal hemorrhage >1 disc area in size and involving the fovea
Time Frame: Baseline through end of study (12 month treatment period)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Number analyzed (Participants) | 513 | 18
Percentage of Participants | 2.9 | 0.0

ADVERSE EVENTS:
Arm/Group | Ranibizumab Non-ANCHOR | Ranibizumab ANCHOR
Serious Adverse Events (participants affected / at risk) | 80/513 | 4/18
Other Adverse Events (participants affected / at risk) | 199/513 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Non-ANCHOR (N=513) | Ranibizumab ANCHOR (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 6 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 5 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Cataract (Fellow eye) (Eye disorders) | 3 | 0
Cataract (Study eye) (Eye disorders) | 1 | 0
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 1 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 2 | 0
Retinal pigment epithelial tear (Study eye) (Eye disorders) | 1 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Cardioactive drug level increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Diabetic coma (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Poor peripheral circulation (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab Non-ANCHOR (N=513) | Ranibizumab ANCHOR (N=18)
Choroidal neovascularisation (Fellow eye) (Eye disorders) | 16 | 2
Choroidal neovascularisation (Study eye) (Eye disorders) | 8 | 2
Conjunctival haemorrhage (Study eye) (Eye disorders) | 28 | 0
Retinal haemorrhage (Fellow eye) (Eye disorders) | 12 | 2
Retinal haemorrhage (Study eye) (Eye disorders) | 35 | 5
Retinal oedema (Study eye) (Eye disorders) | 8 | 2
Visual acuity reduced (Fellow eye) (Eye disorders) | 23 | 1
Visual acuity reduced (Study eye) (Eye disorders) | 94 | 1
Intraocular pressure increased (Study eye) (Investigations) | 36 | 0
Headache (Nervous system disorders) | 13 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.